CLINICAL TRIAL: NCT00913510
Title: Efficacy of Clean Intermittent Self-catheterization in Combination With Anticholinergic Drugs for Treatment of Bladder Dysfunction in Multiple Sclerosis
Brief Title: Efficacy of Clean Intermittent Catheterization (CIC) in Multiple Sclerosis (MS) Patients With Bladder Dysfunction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YA-MSP-0001
Record Dates: First submitted 2009-06-03; First posted 2009-06-04 (Estimated); Results first posted 2014-01-06 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2014-01

CONDITIONS: Bladder Dysfunction; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CIC using LoFric Primo (Experimental): Anticholinergic medication according to clinical practice and investigator´s judgement and start of CIC using LoFric Primo catheters, i.e. Drug + Device.
  Interventions: Device: CIC using LoFric Primo; Drug: Anticholinergic medication
- Anticholinergic medication (Active Comparator): Anticholinergic medication according to clinical practice and investigator´s judgement, i.e. Drug.
  Interventions: Drug: Anticholinergic medication

INTERVENTIONS:
Device: CIC using LoFric Primo — Anticholinergic medication according to clinical practice and investigator´s judgement, either started at screening visit or continued from before study start, and start of CIC using LoFric Primo catheters, i.e. Drug + Device.
  Other Names: LoFric Primo
  Arms: CIC using LoFric Primo
Drug: Anticholinergic medication — Anticholinergic medication according to clinical practice and investigator´s judgement, either started at screening visit or continued from before study start, i.e. Drug.

SUMMARY:
The aims of this prospective, randomized study are:

* To assess the effect of clean intermittent catheterization (CIC)
* To investigate if MS patients will have symptom reduction (urgency, frequency, nocturia and incontinence) when using CIC in combination with anticholinergic drugs
* To identify at what volume of Postvoid Residual (PVR) urine, starting CIC improves bladder control and QoL
* To increase the evidence of CIC, and support clinical guidelines of bladder management in MS patients

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Male and female patients aged 18 years and over
* MS patients that are already currently treated or eligible for treatment with anticholinergic drugs
* Patient with previously confirmed multiple sclerosis according to McDonald Criteria and level of disability less than 6.5 on the Kutzke scale and have been stable for 6 months
* The patient has all or any bladder symptoms; urgency, frequency, incontinence, nocturia, PVR
* The patient has Frequency symptoms > 8 voiding per 24 h
* The patient has PVR > 50 ml, measured at two repetitive bladder scan measurements during the screening phase as well as the randomization visit
* Adequate mobility to lower limbs, sufficient hand function and ability to practice CIC at least three times daily

Exclusion Criteria:

* Pregnancy
* Ongoing symptomatic Urinary Tract Infection (UTI) as judged by investigator
* Involvement in the planning and conduct of the study (applies to both Astra Tech staff or staff at the study site)
* The patient practices CIC prior the study
* The patient has undergone a sphincterectomy
* Progressive "Relapsing- remitting MS" as judged by the investigator
* Severe non-compliance to protocol as judged by the investigator and/or Astra Tech
* The patient is participating in other study that might have an impact on the outcome of this, as judged by investigator
* PVR > 250 ml, measured at two repetitive bladder scan measurements during the screening phase as well as the randomization visit and or if Bladder Voiding Efficiency (BVE) at visit 2 (randomization) is 50% or less than visit 1 (screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clare Fowler, Prof., Principal Investigator — University College, London
Locations (5):
- Belgium (2):
  - Centre Hospitalier Universitaire de Liège Ourthe Ambléve, Esneux
  - UZ Gasthuisberg, Leuven
- St. Hedwig Hospital, Department of Urology, Berlin, Germany
- UMC ST Radboud Nijmegen, Department of Urology, Nijmegen, Netherlands
- University College of London, Institute of Neurology, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study had a screening period between enrolment and randomization. Four (4) of the enroled patients were never randomized due to either withdrawal of consent or not fulfilling inclusion/exclusion criteria at randomization.
Groups:
- CIC Using LoFric Primo: Anticholinergic medication according to clinical practice and investigator´s judgement, either started at screening visit or continued from before study start and start of CIC using LoFric Primo catheters.
- Anticholinergic Medication: Anticholinergic medication according to clinical practice and investigator´s judgement, either started at screening visit or continued from before study start.
Period: Overall Study
Arm/Group | CIC Using LoFric Primo | Anticholinergic Medication
Started | 13 | 7
Completed | 5 | 3
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- CIC Using LoFric Primo: Anticholinergic medication according to clinical practice and investigator´s judgement and start of CIC using LoFric Primo catheters (3-6 times/24h), i.e. Drug + Device
- Total: Total of all reporting groups
Arm/Group | CIC Using LoFric Primo | Anticholinergic Medication | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.15 (12.86) | 51.71 (8.34) | 44.85 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Frequency of Micturition Per Day at 8 Weeks.
Description: Number of micturitions per day was assessed using a patient diary during three days at baseline and after 8 weeks of treatment. The relative change in mean number of micturitions was compared between the groups. The change was calculated as percent change = ((measure at 8 weeks - measure at baseline)/measure at baseline)*100%.
Time Frame: Baseline and 8 weeks after randomization.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | CIC Using LoFric Primo | Anticholinergic Medication
Number analyzed (Participants) | 5 | 3
percent change | -9.09 (27.82) | -6.41 (33.15)
Statistical Analysis 1: Comparison: CIC Using LoFric Primo vs Anticholinergic Medication; H0 : µt = µc versus H1 : µt ≠ µc µt = Exp. relative change of frequency of micturitions per day in test group µc = Exp. relative change of frequency of micturitions per day in control group. Plan was to have 44 evaluable subjects (90% power) but power of the study was reduced by early termination. It cannot be concluded that there is no difference between the treatment groups due to insufficient power; Test type: Superiority or Other; p = 1.0000, Wilcoxon (Mann-Whitney) — The p-value is calculated to the fourth decimal place; Mean Difference (Net) = 2

ADVERSE EVENTS:
Arm/Group | CIC Using LoFric Primo | Anticholinergic Medication
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/7
Other Adverse Events (participants affected / at risk) | 1/13 | 1/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CIC Using LoFric Primo (N=13) | Anticholinergic Medication (N=7)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CIC Using LoFric Primo (N=13) | Anticholinergic Medication (N=7)
Urinary Tract Infection (Renal and urinary disorders) | 1 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days